CLINICAL TRIAL: NCT00297336
Title: An Open-label Observational Safety Study During Administration of Topiramate, for the Prophylaxis of Migraine
Brief Title: An Observational Study Evaluating the Safety of Topiramate for the Prevention of Migraine
Status: Completed | Type: Observational
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Responsible Party: Medical Affairs Director
Other Study IDs: CR002116
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Migraine Disorders
Keywords: Topiramate; Migraine; Headache; Chronic headache; Chronic migraine
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders | interventions — Topiramate

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — 80 patients with diagnosed with migraine

SUMMARY:
A 6-month, observational, post authorization safety study for the collection and evaluation of additional safety data on topiramate as a prophylactic treatment for migraines in adult patients. According to current European and international guidelines the safety and efficacy of drugs will be continuously monitored even after their approval and market circulation.The applicable methods of monitoring include: Observational studies, voluntarily reported adverse events, clinical trials of IV phase and Post Authorization Safety Studies ( PASS). Post Authorization Safety Studies (PASS) during the use of a product are a significant source of information regarding the action of the drug or a therapeutic method under the circumstances of every day clinical practice.

DETAILED DESCRIPTION:
Previous studies have shown that topiramate is effective in preventing migraine headaches. This is a 6-month observational study to evaluate additional safety data of topiramate in the prevention of migraine in adult patients. The study duration is 6-months, with 5 study visits during the study. Administration of topiramate should be according to current Summary of Product Characteristics (SmPC) and daily clinical practice. The decision to prescribe topiramate is decided by the Health Care Professional and it is independent of the protocol. Based on the investigator's judgement, patients who enter the study should fulfill the criteria for administration of prophylactic treatment. In this study a total number of 80 patients with diagnosed migraine according to the criteria of the International Headache Society HIS (Cephalalgia 1998; 8 (Suppl7) :1-98) will participate. Patients who will be enrolled should be either male or female over 18 years of age, fulfilling the above mentioned criteria and who will agree to sign the written informed consent for the anonymous and confidential use of their medical data with their participation in the study. Methods of evaluation include tolerability, laboratory tests, vital signs and Body Weight and Body Mass Index (BMI). Efficacy by assessing migraine attacks, symptomatic medications and Headache Impact Test (HIT-6). Observational study - No investigational drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the IHS (International Headache Society) diagnostic criteria for migraine
* Patients who satisfy the migraine prophylactic medication criteria

Exclusion Criteria:

* Ineligible patient according to the marketed Summary of Product Characteristics of topiramate
* Patient with hypersensitivity to topiramate or to some of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study a total number of 80 patients with diagnosed migraine according to the criteria of the International Headache Society HIS (Cephalalgia 1998; 8 (Suppl7) :1-98) will participate. Patients who will be enrolled should be either male or female over 18 years of age, they should satisfy the migraine prophylactic medication criteria, and will agree to sign the written informed consent for the anonymous and confidential use of their medical data with their participation in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is effectiveness of topiramate based on the frequency of migraine headaches during the monotherapy with topiramate. | Visit 1 and visit 5

SECONDARY OUTCOMES:
Safety of topiramate (number of SAEs, AEs, Laboratory findings) | Visits: 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.